CLINICAL TRIAL: NCT05851859
Title: Randomized Controlled Trial Evaluating the Effectiveness of a Breathing Control Technique on Long COVID Symptoms at the Reunion University Hospital
Brief Title: Evaluation of the Effectiveness of Breathing Control Technique on Long COVID Symptoms at the Reunion University Hospital
Acronym: COCO-Long'Run
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/CHU/35; 2023-A00796-39 (Other: idRCB)
Record Dates: First submitted 2023-05-04; First posted 2023-05-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complementary respiratory training to cardiac coherence (CC) (Experimental): The " intervention " group will benefit from a complementary respiratory training to CC during 6 months in addition to the usual care procedure.
  Interventions: Other: Cardiac coherence
- Usual care procedure in the event of Long COVID (No Intervention): The " control " group will follow a usual care procedure in the event of Long COVID

INTERVENTIONS:
Other: Cardiac coherence — Use of Cardiac coherence (complementary respiratory training) during 6 month
  Arms: Complementary respiratory training to cardiac coherence (CC)

SUMMARY:
Despite the controversy, on October 6, 2021, the World Health Organization (WHO) recognized Long Coronavirus disease (COVID) by officially defining it: " symptoms appeared 3 months after the onset of the primary infection by the Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2), persisting for at least 2 months and which cannot be explained by any other condition ". Long COVID can affects any type of patient and has polymorphic and fluctuating symptoms over time.

The Reunion Island is a French overseas department located in the Indian Ocean accounting more than 860,000 inhabitants. It has recorded since March 11, 2020, nearly 491,825 cases of COVID-19 and 961 deaths of hospitalized patients. Reunion's population is multi-ethnic and younger than the metropolitan France's one. It also has a higher prevalence of obesity and type 2 diabetes, two serious form factors of COVID-19. This specific context makes this island a particular study site for Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) and Long COVID.

In addition, some studies have confirmed the involvement of the autonomic nervous system (ANS) in the symptomatology of Long COVID and demonstrated that patients with a Long COVID present a dysfunction of their ANS which is objectified by a reduced Heart Rate Variability (HRV). The regulation of heart rate by the ANS is strongly favored by respiration. A regular slow and deep breathing training helps to adjust the baroreflex, which connect heart rate, breathing and blood pressure. The result of this training is an induced state called "cardiac coherence" (CC).

The investigator therefore hypothesize that respiratory training to CC could "re-educate" the ANS and durably improve the symptomatology of patients with Long COVID.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18,
* living in Reunion and
* having a diagnosis of Long COVID according to the World Health Organization (WHO) definition will be included in this study.
* These patients must attest to their primary infection with Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) and present a negative antigen test at the time of inclusion.

Exclusion Criteria:

Patients:

* with a chronic or disabling respiratory pathology preventing respiratory training (asthma, Chronic Obstructive Pulmonary Disease (COPD), active tuberculosis, pulmonary sequelae of COVID-19, etc.) practicing or having practiced a regular respiratory control technique (yoga, Cardiac coherence training, etc.) in the last 6 months
* taking a beta-blocker, betamimetic, anti-arrhythmic, morphine, antidepressant treatment (Escitalopram)
* having a pacemaker or severe heart disease
* Current and known pregnancy or breastfeeding woman
* with a cognitive deficit
* under guardianship/curators or under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of a respiratory training to cardiac coherence on the reduction in the symptomatology of patients with Long COVID. | 6 months
  mean score on the Long COVID Symptom Tool (ST) scale Score 0 to 53 / Higher score mean worse outcome

SECONDARY OUTCOMES:
Evaluation of the effectiveness of a respiratory training to cardiac coherence on the decrease of overall symptoms over time | T0, 1 month, 2 months, 3 months, 6 months
  Long COVID Symptom Tool (ST) scale Score 0 to 53 / Higher score mean worse outcome
Evaluation of the effectiveness of a respiratory training to cardiac coherence on the decrease of specifics symptoms : fatigue | 3 months, 6 months
  The 11-item Chalder Fatigue Scale (CFS-11) score 0 to 11 / Higher score mean worse outcome
Evaluation of the effectiveness of a respiratory training to cardiac coherence on the decrease of specifics symptoms : dyspnoea | 3 months, 6 months
  Modified Medical Research Council (MMRC) dyspnoea scale score 0 to 5 / Higher score mean worse outcome
Evaluation of the effectiveness of a respiratory training to cardiac coherence on the decrease of specifics symptoms : Anxiety and Depression | 3 months, 6 months
  Hospital Anxiety and Depression scale (HADS) Score 0 to 42 / Higher score mean worse outcome
Evaluation of the effectiveness of a respiratory training to cardiac coherence on the decrease of specifics symptoms : cognitive disorders | 3 months, 6 months
  Montreal Cognitive Assessment (MoCA) Score 0 to 30 / Higher score mean better outcome
Evaluation of the effectiveness of a respiratory training to cardiac coherence on the decrease of specifics symptoms : Post Traumatic Stress Disorder | 3 months, 6 months
  Posttraumatic Stress Disorder Checklist for Diagnostic and statistical manual of mental disorders, version 5 (PCL-5) Score 0 to 80 / Higher score mean worse outcome
Evaluation of the effectiveness of a respiratory training to CC on the impact of the disease on daily life | T0, 1 month, 2 months, 3 months, 6 months
  Long COVID Impact Tool (IT) scale Score 0 to 60 / Higher score mean worse outcome

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de la Réunion, Saint-Denis
  - CHU de la Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No